CLINICAL TRIAL: NCT06288828
Title: The Efficacy of Aerobic Exercise Training on Autonomic Nervous System and Endothelial Function in Patients with Compensated Cirrhosis: a Parallel, Randomized Controlled Trial
Brief Title: The Efficacy of Aerobic Exercise Training on Autonomic Nervous System and Endothelial Function in Patients with Compensated Cirrhosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Sirinda Kittiprachakul, Principal Investigator, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB0569/66
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Cirrhosis; Aerobic Exercises; Lifestyle Modification; Endothelial Function; Autonomic Nervous System; Autonomic Dysfunction; Heart Rate Variability; Flow Mediated Dilation; Sarcopenia; Physical Activity; Physical Functional Performance; Physical Inactivity
Keywords: Cirrhosis; Autonomic nervous system; Endothelial function; Aerobic exercise
MeSH Terms: conditions — Fibrosis; Primary Dysautonomias; Sarcopenia; Motor Activity; Sedentary Behavior | interventions — Exercise; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Participants in the intervention group will undergo 150 minutes of moderate aerobic exercise per week for 16 weeks, accompanied by a personalized nutritional plan (1.2 grams of protein per kilogram of ideal body weight per day and a calorie intake of 35 kilocalories per kilogram of ideal body weight per day).
  Interventions: Behavioral: Aerobic exercise + Nutrition consultant; Behavioral: Nutrition consultant
- Control group (Other): The control group will solely receive nutritional guidance and maintain their physical inactivity.
  Interventions: Behavioral: Nutrition consultant

INTERVENTIONS:
Behavioral: Aerobic exercise + Nutrition consultant — Participants in the intervention group will engage in 150 minutes of moderate aerobic exercise weekly for 16 weeks, primarily brisk walking or jogging.
  For the initial four weeks, they will visit the hospital weekly for guidance and participate in home-based exercise following a protocol totaling 150 minutes of moderate aerobic exercise in the form of brisk walking or jogging. Healthcare professionals will help adjust exercise intensity based on heart rate (60-80% of maximum) and perceived exertion (RPE 12-15), while monitoring vital signs and adverse events.
  After, they will transition to a home exercise program for twelve weeks, recording exercise details in a logbook. Weekly follow-up calls will ensure adherence and monitor adverse events.
  They will be provided with nutritional recommendations by a dietitian, the same as the control group.
  Other Names: Exercise group; Active group
  Arms: Exercise group
Behavioral: Nutrition consultant — Participants will maintain their physical activity at the same level as before enrolling in the study.
  However, they will be provided with nutritional recommendations by a dietitian, which include 1.2 grams of protein per kilogram of ideal body weight daily and a calorie intake of 35 kilocalories per kilogram of ideal body weight per day. To assess adherence and make necessary adjustments, participants will complete a 3-day food record at the beginning of the study, at week 8, and at the end of the study at week 16. If participants encounter difficulties adhering to the recommended nutritional intake, the dietitian will provide additional guidance to help them meet the requirements.
  Other Names: diet

SUMMARY:
The goal of this clinical trial is to explore the impact of a 16-week aerobic exercise regimen on the autonomic nervous system and endothelial function in patients with compensated cirrhosis who have physical inactivity. The primary research question is:

1) What effect does 16 weeks of aerobic exercise have on changes in the autonomic nervous system and endothelial function in cirrhotic patients?

Additionally, the secondary research questions are:

1. How does a 16-week aerobic exercise program influence changes in muscle mass, muscle strength, and physical performance in cirrhotic patients?
2. Is there a correlation between muscle mass and parameters of the autonomic nervous system in cirrhotic patients?

Participants in the intervention group will undergo 150 minutes of moderate aerobic exercise per week for 16 weeks, accompanied by a personalized nutritional plan (1.2 grams of protein per kilogram of ideal body weight per day and a calorie intake of 35 kilocalories per kilogram of ideal body weight per day). The control group will solely receive nutritional guidance and maintain their physical inactivity. The researchers will compare outcomes between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of cirrhosis is confirmed either through liver biopsy ,and/or compatible features on ultrasonography/ computer tomography or magnetic resonance imaging.
* The age range is between 45 and 75 years.
* Participants are classified as Child Pugh score class A.
* Participants report a physical inactivity, defined as engaging in physical activity for less than 150 minutes of moderate-intensity physical activity per week, or less than 75 minutes of vigorous-intensity physical activity per week, or an equivalent combination of both.

Exclusion Criteria:

* Active hepatocellular carcinoma (HCC) or remission of HCC within the past 3 months.
* Untreated large esophageal varices (EV) greater than F2 or history of upper gastrointestinal bleeding from portal hypertension or gastric varices.
* Active or history of hepatic encephalopathy (HE).
* Inpatient hospitalization for any reason or discharge from the hospital within the past 3 months.
* Complete portal vein thrombosis.
* Transjugular intrahepatic portosystemic shunt.
* Contraindications to exercise, such as recent myocardial infarction, unstable angina, electrocardiography changes within the past 24 hours, complete heart block, acute congestive heart failure, uncontrolled hypertension, hemoglobin level less than 11 g/dL, platelet count less than 50,000 cells/mm 3 .
* End-stage renal disease without dialysis.
* Severe orthopedic problems that limit the ability to exercise.
* Inability to communicate with the research team via telemedicine system.
* Body mass index (BMI) exceeding 35 kg/m 2 .
* On alpha or beta-blocker

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1.Autonomic function test: Heart rate variability (HRV), Ewing autonomic battery test | The study duration will span from enrollment through treatment completion at 16 weeks or within 2 weeks after the end of the study
  HRV:
  Time-domain: SDNN (milliseconds), SD of delta NN (milliseconds), o RMSSD, Mean spectrum NN (milliseconds), NN50 (%) Frequency-domain: Very Low-Frequency (VLF) Power, Low-Frequency (LF) Power, High-Frequency (HF) Power , LF/HF Ratio
Endothelial function test: Flow mediated dilation (FMD) in % FMD change | The study duration will span from enrollment through treatment completion at 16 weeksor within 2 weeks after the end of the study

SECONDARY OUTCOMES:
Physical function | The study duration will span from enrollment through treatment completion at 16 weeks, plus or minus 2 weeks".
  6-minute walk test (minute)
Muscle mass change | The study duration will span from enrollment through treatment completion at 16 weeks, or within 2 weeks after the end of the study
  Lean appendicular mass (kg) from Dual energy X-ray absorptiometry (DXA)
Muscle strength change | The study duration will span from enrollment through treatment completion at 16 weeks, or within 2 weeks after the end of the study
  Handgrip strength (kg) from dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text,tables,figures, and appendices) will be provided with anyone who wishes to access the data.
  Study Protocol will also be provided with anyone who wishes to access the data.
  Information regarding submitting proposals and accessing data may be found at https://rehabmed.md.chula.ac.th/research/.
Supporting Information: Study Protocol
Time Frame: The data will be begin 9 months and end 36 months following article publication.
Access Criteria: Share via E-mail on request Contact: sirinda.ning@gmail.com